CLINICAL TRIAL: NCT06221865
Title: Study of the Correlation Between Post-traumatic Stress Disorder and Paradoxical Sleep Behavior Disorder
Acronym: TRAUMA-TCSP
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2023 FANTINI
Record Dates: First submitted 2024-01-08; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2023-12

CONDITIONS: Post Traumatic Stress Disorder; Sleep Disorder
Keywords: Post Traumatic Stress Disorder; Sleep disorders; Rapid eye movement sleep behavior disorder; Data Correlation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sleep Wake Disorders; REM Sleep Behavior Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Post-Traumatic Stress Disorder is a psychiatric disorder that occurs after a traumatic event and is estimated to affect 5 to 12% of the general population. Around 70% of patients suffering from this disorder report sleep disorders (sleep apnea, insomnia, recurring nightmares, etc.).

There are specific sleep disorders called Rapid Eye Movement (REM) sleep behavior disorders which correspond to nocturnal restlessness with sometimes violent behavior, often associated with intense dreams during a phase of sleep called REM sleep. These disorders are more frequently found in patients suffering from post-traumatic stress, such as veterans.

However, the physiopathological link between these two disorders is poorly understood and studies on this subject are few in number. Through this study, the investigators wish to demonstrate whether there is a correlation between the severity of Post-Traumatic Stress Disorder and that of Rapid Eye Movement sleep behavior disorder.

The main objective is to study the relationship between the severity of Post Traumatic Stress Disorder (PTSD) and the Rapid Eye Movement (REM) Sleep Behavior Disorder.

This is an observational prospective study based on 4 questionnaires relating to the sleep (PSQI), the severity of the Rapid Eye Movement (REM) Sleep Behavior Disorder (REM RBDSQ, IRBD-SSS) and the severity of the Post-Traumatic Stress Disorder (PCL-5).

DETAILED DESCRIPTION:
Type of study: observational prospective study

Study duration : 40 min, one visit at D0 (inclusion isit)

Number of center: 1 (Clermont Ferrand)

Patients: 60 patients suffering from type 1 Post-traumatic Stress Disorder .

Patients will be selected during their consultation, at the CUMP (Medico-Psychological Emergency Cell) of the hospital of Clermont-Ferrand. If patients accept to participate to this study, demographic and clinical data (age, sex, current treatments, medical and surgical history) will be collected. Then, they will complete 4 questionnaires :

* the Rapid Eye Movement Behavior Disorder Screening Questionnaire (REM RBDSQ)
* the Rapid Eye Movement Behavior Disorder symptom severity scale score (IRBDSSS)
* the quality of sleep inventory (PSQI)
* the Posttraumatic Stress Disorder Checklist for DSM-5 (PCL 5)

ELIGIBILITY:
Inclusion Criteria:

* Adult patient aged 18 to 50 years.
* French speaking.
* Having a diagnosis of type I Posttraumatic Stress Disorder according to DSM 5.

Exclusion Criteria:

* Presence of acute mental illnesses in the process of decompensation.
* Presence of a Central Nervous System disorder (e.g. neurodegenerative diseases, Stroke, Multiple Sclerosis (MS), Narcolepsy, etc.)
* Patient under guardianship, curatorship, or legal protection.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 60 patients suffering from type 1 Post-traumatic Stress Disorder (PTSD) will be included in this study. They will be selected during their consultation at the CUMP (Cellule d'Urgence Medico Psychologique) of the hospital of Clermont-Ferrand.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Severity of the Posttraumatic Stress Disorder score | Day 0
  This self-questionnaire is completed by the patient during the inclusion visit
Severity of the Rapid Eye Movement Behavior Disorder symptom score | Day 0
  This self-questionnaire is completed by the patient during the inclusion visit

SECONDARY OUTCOMES:
The Rapid Eye Movement Behavior Disorder Screening Questionnaire score | Day 0
  This self-questionnaire is completed by the patient during the inclusion visit
The quality of sleep inventory score | Day 0
  This self-questionnaire is completed by the patient during the inclusion visit

CONTACTS AND LOCATIONS:
Overall Officials: Livia Fantini, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France